CLINICAL TRIAL: NCT06644768
Title: A Multicenter, Randomized, Open-Label, Phase 1b/2 Trial Of Valemetostat Tosylate Plus Pembrolizumab Vs Pembrolizumab Alone in Participants With Advanced or Metastatic Non-Small Cell Lung Cancer Whose Tumors Express PD-L1 With Tumor Proportion Score ≥50% Without Actionable Genomic Alterations
Brief Title: A Study of Valemetostat Tosylate Plus Pembrolizumab Versus Pembrolizumab Alone in First-Line NSCLC Without Actionable Genomic Alterations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS3201-330; MK-3475-F85 (Other: Merck Sharp & Dohme LLC); KEYNOTE-F85 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2024-10-01; First posted 2024-10-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer; Lung Cancer
Keywords: NSCLC; Tumor; pembrolizumab; valemetostat tosylate; DS-3201b; Immune checkpoint inhibitor; Programmed Cell Death 1 Ligand 1; MK-3475
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1b: Pembrolizumab + Valemetostat Tosylate (Experimental): Participants will be provided with pembrolizumab at standard dose of 200 mg intravenously (IV) Q3W, and valemetostat will be provided per a dose escalation schedule, with an initial starting dose of 150 mg by mouth once daily.
  Interventions: Drug: valemetostat tosylate; Drug: pembrolizumab
- Phase 2: Pembrolizumab + Valemetostat Tosylate (Experimental): Participants will be provided with pembrolizumab at standard dose of 200 mg IV Q3W, and valemetostat will be provided per recommended phase 2 dose (RP2D)
  Interventions: Drug: valemetostat tosylate; Drug: pembrolizumab
- Phase 2: Pembrolizumab (Active Comparator): Participants will be provided with pembrolizumab at standard dose of 200 mg IV Q3W
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: valemetostat tosylate — Valemetostat will be administered orally once daily until RP2D of valemetostat is determined.
  Other Names: DS-3201b; valemetostat
  Arms: Phase 1b: Pembrolizumab + Valemetostat Tosylate; Phase 2: Pembrolizumab + Valemetostat Tosylate
Drug: pembrolizumab — One IV infusion Q3W on D1 of each 21-day cycle for a maximum of 35 cycles.
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
This study will compare Valemetostat Tosylate Plus Pembrolizumab vs Pembrolizumab Alone in First-line NSCLC Without Actionable Genomic Alterations

DETAILED DESCRIPTION:
This trial will evaluate the safety and efficacy of valemetostat tosylate (DS-3201b) in combination with fixed-dose pembrolizumab versus pembrolizumab alone in participants with advanced or metastatic NSCLC without actionable genomic alterations, whose tumor has PD-L1 TPS ≥50%, and who have not received prior systemic therapy for advanced or metastatic NSCLC. The trial will be in 2 phases, dose escalation and dose expansion phases.

ELIGIBILITY:
Key Inclusion Criteria:

1. Has signed and dated the ICF, prior to the start of any trial-specific qualification procedures.
2. Is an adult ≥18 years of age or the minimum legal age (whichever is greater) at the time of informed consent. (Follow local regulatory requirements if the legal age of adult voluntary consent for trial participation is >18 years old).
3. Has histologically documented NSCLC that meets all of the following criteria:

   1. Has no prior systemic therapy for advanced or metastatic disease.
   2. Has Stage IIIB or IIIC disease and is not a candidate for surgical resection or definitive chemoradiation, or Stage IV NSCLC disease at the time of enrollment/randomization (based on the American Joint Committee on Cancer, Eighth Edition). Participants with early-stage NSCLC who have relapsed should be restaged during Screening to ensure their eligibility for the trial.
   3. Has documented negative test results for EGFR, ALK, and ROS1 actionable genomic alterations based on analysis of tumor tissue. If test results for EGFR, ALK, and ROS1 are not available, participants are required to undergo testing performed locally for these genomic alterations.

      Participants with squamous NSCLC are only required to undergo EGFR, ALK, and ROS1 testing if they have no history of tobacco smoking or were diagnosed with NSCLC at <40 years of age.
   4. Has no known actionable genomic alterations in NTRK, BRAF, RET, MET, or other actionable oncogenic drivers with locally approved therapies (testing for genomic alterations besides EGFR, ALK, and ROS1 is not required prior to enrollment/randomization). Participants whose tumors harbor KRAS mutations are eligible for the trial.
4. Has measurable disease on CT or MRI based on local imaging assessment using RECIST v1.1
5. Has a tumor expressing PD-L1 TPS ≥50% as determined by local testing using 22C3 pharmDx PD-L1 IHC assay. In regions where PD-L1 (TPS ≥50%) testing by 22C3 pharmDx is not considered SOC, PD-L1 expression levels will be determined by central testing (minimum of 6 slides).
6. Has provided a formalin-fixed tumor tissue sample for the assessment of biomarkers. This tissue requirement is in addition to the tissue required for PD-L1 testing for tissue screening purposes. If a documented law or regulation prohibits (or does not approve) sample collection, then such sample will not be collected.
7. Has an ECOG PS of 0 or 1 at Screening.

Key Exclusion Criteria

1. Has received prior treatment with any of the following, including in the adjuvant/neoadjuvant setting:

   1. Any anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX40, or CD137).
   2. Has previously been treated with any enhancer of zeste homolog inhibitors.
2. Participants who received adjuvant or neoadjuvant therapy other than those listed in the exclusion criterion above are eligible if the adjuvant/neoadjuvant therapy was completed at least 6 months prior to the current diagnosis of advanced or metastatic disease.
3. Has received a live vaccine or live attenuated vaccine within 30 days prior to the first dose of trial intervention. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccines. Note: Administration of killed vaccines is allowed.
4. Has an active, known, or suspected autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of systemic disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.

   Inhaled, intranasal, intraocular, intra-articular, or topical steroids and adrenal replacement steroids are permitted in the absence of active autoimmune disease.
5. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (at doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial intervention. Note: Short-course systemic corticosteroids (eg, prevention of/treatment for transfusion reaction) or steroid use for a noncancer indication (eg, adrenal replacement) is permissible.
6. Has a known active or untreated CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate, provided they are radiologically stable (ie, without evidence of progression) for at least 4 weeks by repeat imaging (note: repeat imaging should be performed during trial screening), clinically stable, and without requirement of steroid treatment for at least 14 days before the first dose of trial intervention. Note: A CT scan or MRI scan of the brain at Baseline is required for all participants. For participants in whom CNS metastases are first discovered at Screening, the treating investigator should delay trial intervention to complete any necessary treatment followed by a proper washout period and document the stability of CNS metastases with repeat imaging at least 4 weeks later (in which case repetition of all screening activities may be required).
7. Has uncontrolled or significant cardiovascular disease, including the following:

   1. Mean QT interval corrected for heart rate using Fridericia's formula >470 ms (based on the average of screening triplicate 12-lead ECG determinations)
   2. Myocardial infarction within 6 months prior to Screening
   3. Uncontrolled angina pectoris within 6 months prior to Screening
   4. New York Heart Association Class 3 or 4 congestive heart failure
   5. Uncontrolled hypertension (resting systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg)
8. Has a history of (noninfectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
9. Has a history of radiation pneumonitis.
10. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Number of Participants with Dose-Limiting Toxicities | From day of first dose on Day 1 to Day 21 in Cycle 1 (21 days), or before the administration of Cycle 2, up to 24 days
  Total number of participants with A Dose-Limiting Toxicity (DLT) at each dose level of valemetostat in combination with pembrolizumab per National Cancer Institute - Common Terminology Criteria for Adverse Events version 5.0.
Phase 1b: Number of Participants with Treatment-Emergent Adverse Events | From date of first dose to 30 days after last dose, up to approximately 31 months
  Incidence of TEAEs, Grade 3 or 4 TEAEs, deaths, TESAEs, TEAEs leading to dose modifications (including interruption, reduction, and discontinuation), and AESIs using the National Cancer Institute - Common Terminology Criteria for Adverse Events version 5.0
Phase 2: Progression-Free Survival by BICR | From date of randomization to the date of radiographic disease progression, or death from any cause, whichever occurs first, up to approximately 31 months
  PFS is the time from the date of randomization to the date of radiographic disease progression as assessed by blinded independent central review (BICR) per RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Phase 2: Objective Response Rate | From date of randomization to the date of radiographic disease progression, or death from any cause, whichever occurs first, up to approximately 31 months
  Objective Response Rate (ORR) is the proportion of participants with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) assessed by BICR.
Phase 2: Duration of Response | From date of randomization to the date of radiographic disease progression, or death from any cause, whichever occurs first, up to approximately 31 months
  Duration of Response (DoR) is the time from the date of first documentation of objective tumor response (CR or PR) that is subsequently confirmed to the date of the first documentation of objective tumor progression or to death from any cause, whichever occurs first, assessed by BICR.
Phase 2: Disease Control Rate | From date of randomization up to approximately 31 months
  Disease control rate (DCR) is the proportion of participants who achieved a BOR of confirmed CR, confirmed PR, or stable disease (SD), assessed by BICR.
Phase 2: Overall Survival | From date of randomization the date of death from any cause, up to approximately 31 months
  Overall Survival (OS ) is the time from the date of randomization to the date of death from any cause.
Phase 2: Progression-Free Survival by Investigator | From date of randomization to the date of radiographic disease progression, or death from any cause, whichever occurs first, up to approximately 31 months
  PFS is the time from the date of randomization to the date of radiographic disease progression as assessed by the investigator per RECIST v1.1 or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (45):
- United States (12):
  - University of California San Diego (Ucsd)-Moores Cancer Center, La Jolla, California
  - California Research Institute, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Mayo Clinic Hospital, Jacksonville, Florida
  - BRCR Global, Plantation, Florida
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Virginia Cancer Specialist, Fairfax, Virginia
- Argentina (7):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Sanatorio Allende, Córdoba
  - Fundacion Ars Medica, N Salvador de Jujuy
  - Centro de Investigacion Pergamino Sa, Pergamino
  - Instituto Medico de La Fundacion Estudios Clinicos, Rosario
  - Clinica Viedma S.A., Viedma
- Brazil (7):
  - Centro de Pesquisas Clinica Reichow, Blumenau
  - Clínica de Neoplasias Litoral Ltda., ItajaĂ-
  - CINPAM Centro Integrado De Pesquisa Da Amazonia, Manaus
  - Liga Norte-Rio-Grandense Contra o Câncer, Natal
  - Hospital Nossa Senhora da Conceicao, Porto Alegre
  - Cepho - Centro de Estudos E Pesquisas de Hematologia E Oncologia, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto, Sao Jose Rio Preto
- China (10):
  - Jilin Cancer Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - Chengdu Shang Jin Nan Fu Hospital, Chengdu
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiamusi Cancer Hospital, Jiamusi
  - Shanghai East Hospital, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tiyuan
  - Henan Cancer Hospital, Zhengzhou
- Japan (5):
  - Kyushu University Hospital, Fukuoka
  - National Cancer Center Hospital East, Kashiwa
  - Cancer Institute Hospital of JFCR, Kōtoku
  - NHO Nagoya Medical Center, Nagoya
  - Kitasato University Hospital, Sagamihara-shi
- South Korea (4):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, St. Vincent'S Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/